CLINICAL TRIAL: NCT06514794
Title: A Phase 2 Study of WU-CART-007, an Anti-CD7 Allogeneic CAR-T Cell Therapy in Patients With Relapsed/Refractory Cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma (T-RRex)
Brief Title: A Phase 2 Study of WU-CART-007, an Anti-CD7 Allogeneic CAR-T Cell Therapy in T-Cell Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma (T-RRex)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wugen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WUC007-03
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: CAR-T Therapy
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: The study is divided into 2 cohorts:
  Relapsed/Refractory (R/R) Cohort will evaluate patients with relapsed or refractory disease
  Minimal Residual Disease (MRD) Positive Cohort will evaluate patients in complete remission with MRD positive disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- WU-CART-007 (Experimental): A CD7-directed chimeric antigen receptor (CAR) T-cell product.
  Lymphodepletion
  Interventions: Biological: WU-CART-007

INTERVENTIONS:
Biological: WU-CART-007 — A single IV infusion of WU-CART-007

SUMMARY:
The T-RRex study evaluates the efficacy of WU-CART-007 for patients with Relapsed/Refractory (R/R) T-Cell Acute Lymphoblastic Leukemia (T-ALL)/Lymphoblastic Lymphoma (LBL) and to WU-CART-007 as a therapy to induce complete Minimum Residual Disease (MRD) negative response

DETAILED DESCRIPTION:
This is a Phase 2, single-arm, multi-center, open label study in patients with R/R T-ALL/LBL and T-ALL/LBL in remission but remaining MRD positive.

ELIGIBILITY:
Key Inclusion Criteria:

* Disease Criteria: Evidence of T-ALL or T-LBL, as defined by World Health Organization (WHO) classification, and either relapse/refractory or MRD positive
* Age: Lower age limit of ≥ 1 year; adequate organ function
* Eastern Cooperative Oncology Group (ECOG)/Karnofsky Performance Status 0 or 1/70 and above at Screening.

Key Exclusion Criteria:

* Prior treatment with any anti-CD7 therapy.
* Patients with decompensated hemolytic anemia.
* Presence of Grade 2 to 4 acute or extensive chronic GvHD requiring systemic immunosuppression. Grade 1 GvHD not requiring immunosuppression or Grade 2 skin GvHD if treated with topical therapy only are acceptable.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
R/R Cohort - Composite Complete Response Rate | 24 months
  CRc is defined as proportion of patients that achieve a complete remission (CR) + CR with incomplete hematologic recovery (CRi)
MRD Pos Cohort - Response Rate | 24 months
  Defined as the efficacy of WU-CART-007 to induce complete MRD negative response

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Thomas, MD, Study Director — Wugen, Inc.
Locations (10):
- United States (8):
  - City of Hope, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Tampa, Florida
  - Washington University Saint Louis, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Peter Mac Callum Cancer Institute, Melbourne, Victoria
  - Royal Children's Melbourne, Melbourne, Victoria